CLINICAL TRIAL: NCT04923529
Title: Phase II Trial of TAS-102 in Patients With Advanced, Refractory Pancreatic Adenocarcinoma
Brief Title: TAS-102 in Patients With Advanced, Refractory Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Chi-Leung Chiang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-711
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pancreas Cancer
Keywords: Pancreatic Adenocarcinoma; TAS-102
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-102 (Experimental): Single group assignment of TAS-102 in Patients with Advanced, Refractory Pancreatic Adenocarcinoma
  Interventions: Drug: TAS 102

INTERVENTIONS:
Drug: TAS 102 — Days 1 through 5: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 1 of each cycle and the last dose administered in the evening of Day 5.
  Days 6 through 7: Recovery
  Days 8 through 12: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 8 of each cycle and the last dose administered in the evening of Day 12.
  Days 13 through 28: Recovery

SUMMARY:
This is a prospective phase II, single arm clinical trial conducted in Queen Mary Hospital (Hong Kong) assessing the efficacy and safety of TAS-102 in advanced or metastatic pancreatic cancer patients.

DETAILED DESCRIPTION:
All the patients must be registered with the Investigator(s) prior to initiation of treatment. The registration desk will confirm all eligibility criteria and obtain essential information (including patient number).

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmed advanced or metastatic pancreatic cancer
2. Measurable disease according to the RECIST criteria (version 1.1) for the evaluation of measurable disease
3. Documented progression after one or more lines of systemic chemotherapy

   1. For the treatment of advanced or metastatic disease
   2. Within 6 months after completion of neo-adjuvant therapy or adjuvant therapy
4. Age ≥ 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance 0-1
6. Written informed consent obtained for clinical trial participation and providing archival tumor tissue, if available
7. Females of childbearing potential or non-sterilized male who are sexually active must use a highly effective method of contraception
8. Females of childbearing potential must have negative serum or urine pregnancy test
9. Have life expectancy ≥ 3 months
10. Adequate organ function as defined as:

    1. Hemoglobin value of ≥9.0 g/dL.
    2. Absolute neutrophil count of ≥1,500/mm3 (IU: ≥1.5 × 10^9/L).
    3. Platelet count ≥100,000/mm3 (IU: ≥100 × 10^9/L).
    4. Total serum bilirubin of ≤1.5 mg/dL (except for Grade 1 hyperbilirubinemia due solely to a medical diagnosis of Gilbert's syndrome).
    5. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤3.0 × upper limit of normal (ULN); if liver function abnormalities are due to underlying liver metastasis, AST and ALT ≤5 × ULN.
    6. Serum creatinine of ≤1.5 mg/dL

Exclusion Criteria:

1. Has disease that is suitable for local therapy administrated with curative intent
2. Has a serious illness or medical condition(s) including, but not limited to the following:

   1. Other concurrently active malignancies excluding malignancies that are disease free for more than 5 years or carcinoma-in-situ deemed cured by adequate treatment.
   2. Known brain metastasis or leptomeningeal metastasis.
   3. Active infection (i.e. body temperature ≥38°C due to infection).
   4. Ascites, pleural effusion or pericardial fluid requiring drainage in last 4 weeks.
   5. Intestinal obstruction, pulmonary fibrosis, renal failure, liver failure, or cerebrovascular disorder.
   6. Uncontrolled diabetes.
   7. Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure New York Heart Association (NYHA) class III or IV
   8. Gastrointestinal hemorrhage.
   9. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or hepatitis B or C.
   10. Patients with autoimmune disorders or history of organ transplantation who require immunosuppressive therapy.
   11. Psychiatric disease that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results.
3. Has had treatment with any of the following within the specified time frame prior to study drug administration:

   1. Major surgery within prior 4 weeks.
   2. Any systemic therapy within prior 2 weeks.
   3. Any radiation within prior 2 weeks.
   4. Any investigational agent received within prior 4 weeks.
4. Untreated active hepatitis B or hepatitis C infections.
5. Has received TAS-102.
6. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation and platinum-induced neurotoxicity).
7. Is a pregnant or lactating female.
8. Is inappropriate for entry into this study in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
16-week progression-free survival (PFS) rate | From the date of informed consent to radiographically documented progression according to RECIST 1.1, assessed up to 16 weeks
  The percentage of study population alive and without progression (according to RECIST 1.1) at 16 weeks from the date of informed consent

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | from the date of informed consent to radiographically documented progression according to RECIST 1.1 or death from any cause, whichever occurs first, assessed up to 3 years
  PFS is measured from the date of informed consent to radiographically documented progression according to RECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow up will be censored at the date of their last radiographic assessment.
Time to progression (TTP) | from the date of informed consent to radiographically documented progression according to RECIST 1.1, assessed up to 3 years
  TTP is measured from the date of informed consent to radiographically documented progression according to RECIST 1.1. Participants death and without disease progression, alive without disease progression, or lost to follow-up will be censored at the date of their last radiographic assessment
Overall survival (OS) | from the date of informed consent to the date of death from any cause, assessed up to 5 years
  OS is measured from date of informed consent to the date of death from any cause. Participants alive or lost to follow-up will be censored at the date of their last radiographic assessment
Objective response rate (ORR) | From the date of first study treatment to radiographically documented complete response or partial response according to RECIST 1.1, assessed up to 3 years
  The percentage of patients with radiologically complete or partial response as determined by the Investigator according to RECIST version 1.1.
Disease control rate (DCR) | from the date of first study treatment to radiographically documented complete response, partial response, or stable disease according to RECIST 1.1, assessed up to 3 years
  The percentage of patients with radiologically complete response, partial response, or stable disease as determined by the Investigators according to RECIST version 1.1
Duration of response (DoR) | from the date of documentation of tumor response to radiographically documented progression according to RECIST 1.1, assessed up to 3 years
  DoR is the time from documentation of tumor response to radiographically documented disease progression
Time to deterioration of ECOG performance status | from the date of informed consent to the first date on which ECOG performance status scores 2 or higher, assessed up to 3 years
  Time from date of informed consent until the first date on which ECOG performance status score of 2 or higher was recorded
Time to deterioration of quality of life | from the date of informed consent to recorded decrease of 10 points or more in EORTC QLQ-C30 assessment, assessed up to 3 years
  Decrease from baseline of 10 points or more on the EORTC QLQ-C30 maintained for two consecutive assessments or a decrease of 10 points or more in one assessment followed by death from any cause within 3 weeks
Incidence of Study-Related Adverse Events [Safety and Tolerability] | from the date of first study treatment to occurrence of study-related adverse events based on NCI-CTCAE 5, assessed up to 3 years
  Incidence, nature, and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE 5)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Leung Chiang, FRCR, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, HKU, Hong Kong, Hong Kong

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328
- [Background] Oettle H, Riess H, Stieler JM, Heil G, Schwaner I, Seraphin J, Gorner M, Molle M, Greten TF, Lakner V, Bischoff S, Sinn M, Dorken B, Pelzer U. Second-line oxaliplatin, folinic acid, and fluorouracil versus folinic acid and fluorouracil alone for gemcitabine-refractory pancreatic cancer: outcomes from the CONKO-003 trial. J Clin Oncol. 2014 Aug 10;32(23):2423-9. doi: 10.1200/JCO.2013.53.6995. Epub 2014 Jun 30. PMID 24982456
- [Background] Gill S, Ko YJ, Cripps C, Beaudoin A, Dhesy-Thind S, Zulfiqar M, Zalewski P, Do T, Cano P, Lam WYH, Dowden S, Grassin H, Stewart J, Moore M. PANCREOX: A Randomized Phase III Study of Fluorouracil/Leucovorin With or Without Oxaliplatin for Second-Line Advanced Pancreatic Cancer in Patients Who Have Received Gemcitabine-Based Chemotherapy. J Clin Oncol. 2016 Nov 10;34(32):3914-3920. doi: 10.1200/JCO.2016.68.5776. Epub 2016 Sep 30. PMID 27621395
- [Background] Ioka T, Komatsu Y, Mizuno N, Tsuji A, Ohkawa S, Tanaka M, Iguchi H, Ishiguro A, Kitano M, Satoh T, Yamaguchi T, Takeda K, Kida M, Eguchi K, Ito T, Munakata M, Itoi T, Furuse J, Hamada C, Sakata Y. Randomised phase II trial of irinotecan plus S-1 in patients with gemcitabine-refractory pancreatic cancer. Br J Cancer. 2017 Feb 14;116(4):464-471. doi: 10.1038/bjc.2016.436. Epub 2017 Jan 12. PMID 28081543
- [Background] Ueno M, Okusaka T, Omuro Y, Isayama H, Fukutomi A, Ikeda M, Mizuno N, Fukuzawa K, Furukawa M, Iguchi H, Sugimori K, Furuse J, Shimada K, Ioka T, Nakamori S, Baba H, Komatsu Y, Takeuchi M, Hyodo I, Boku N. A randomized phase II study of S-1 plus oral leucovorin versus S-1 monotherapy in patients with gemcitabine-refractory advanced pancreatic cancer. Ann Oncol. 2016 Mar;27(3):502-8. doi: 10.1093/annonc/mdv603. Epub 2015 Dec 17. PMID 26681680
- [Background] Ohkawa S, Okusaka T, Isayama H, Fukutomi A, Yamaguchi K, Ikeda M, Funakoshi A, Nagase M, Hamamoto Y, Nakamori S, Tsuchiya Y, Baba H, Ishii H, Omuro Y, Sho M, Matsumoto S, Yamada N, Yanagimoto H, Unno M, Ichikawa Y, Takahashi S, Watanabe G, Wakabayashi G, Egawa N, Tsuda M, Hosotani R, Hamada C, Hyodo I. Randomised phase II trial of S-1 plus oxaliplatin vs S-1 in patients with gemcitabine-refractory pancreatic cancer. Br J Cancer. 2015 Apr 28;112(9):1428-34. doi: 10.1038/bjc.2015.103. Epub 2015 Apr 16. PMID 25880004
- [Background] Ge F, Xu N, Bai Y, Ba Y, Zhang Y, Li F, Xu H, Jia R, Wang Y, Lin L, Xu J. S-1 as monotherapy or in combination with leucovorin as second-line treatment in gemcitabine-refractory advanced pancreatic cancer: a randomized, open-label, multicenter, phase II study. Oncologist. 2014 Nov;19(11):1133-4. doi: 10.1634/theoncologist.2014-0223. Epub 2014 Oct 1. PMID 25273077
- [Background] Hosein PJ, de Lima Lopes G Jr, Pastorini VH, Gomez C, Macintyre J, Zayas G, Reis I, Montero AJ, Merchan JR, Rocha Lima CM. A phase II trial of nab-Paclitaxel as second-line therapy in patients with advanced pancreatic cancer. Am J Clin Oncol. 2013 Apr;36(2):151-6. doi: 10.1097/COC.0b013e3182436e8c. PMID 22307213
- [Background] Ko AH, Tempero MA, Shan YS, Su WC, Lin YL, Dito E, Ong A, Wang YW, Yeh CG, Chen LT. A multinational phase 2 study of nanoliposomal irinotecan sucrosofate (PEP02, MM-398) for patients with gemcitabine-refractory metastatic pancreatic cancer. Br J Cancer. 2013 Aug 20;109(4):920-5. doi: 10.1038/bjc.2013.408. Epub 2013 Jul 23. PMID 23880820
- [Background] Sudo K, Yamaguchi T, Nakamura K, Denda T, Hara T, Ishihara T, Yokosuka O. Phase II study of S-1 in patients with gemcitabine-resistant advanced pancreatic cancer. Cancer Chemother Pharmacol. 2011 Feb;67(2):249-54. doi: 10.1007/s00280-010-1311-3. Epub 2010 Mar 30. PMID 20352216
- [Background] Yi SY, Park YS, Kim HS, Jun HJ, Kim KH, Chang MH, Park MJ, Uhm JE, Lee J, Park SH, Park JO, Lee JK, Lee KT, Lim HY, Kang WK. Irinotecan monotherapy as second-line treatment in advanced pancreatic cancer. Cancer Chemother Pharmacol. 2009 May;63(6):1141-5. doi: 10.1007/s00280-008-0839-y. Epub 2008 Oct 7. PMID 18839175
- [Background] Morizane C, Okusaka T, Furuse J, Ishii H, Ueno H, Ikeda M, Nakachi K, Najima M, Ogura T, Suzuki E. A phase II study of S-1 in gemcitabine-refractory metastatic pancreatic cancer. Cancer Chemother Pharmacol. 2009 Jan;63(2):313-9. doi: 10.1007/s00280-008-0741-7. Epub 2008 Apr 9. PMID 18398614
- [Background] Boeck S, Wilkowski R, Bruns CJ, Issels RD, Schulz C, Moosmann N, Laessig D, Haas M, Golf A, Heinemann V. Oral capecitabine in gemcitabine-pretreated patients with advanced pancreatic cancer. Oncology. 2007;73(3-4):221-7. doi: 10.1159/000127413. Epub 2008 Apr 17. PMID 18424886
- [Background] Boeck S, Weigang-Kohler K, Fuchs M, Kettner E, Quietzsch D, Trojan J, Stotzer O, Zeuzem S, Lordick F, Kohne CH, Kroning H, Steinmetz T, Depenbrock H, Heinemann V. Second-line chemotherapy with pemetrexed after gemcitabine failure in patients with advanced pancreatic cancer: a multicenter phase II trial. Ann Oncol. 2007 Apr;18(4):745-51. doi: 10.1093/annonc/mdl463. Epub 2007 Jan 17. PMID 17229775
- [Background] Androulakis N, Syrigos K, Polyzos A, Aravantinos G, Stathopoulos GP, Ziras N, Mallas K, Vamvakas L, Georgoulis V; Hellenic Oncology Research Group. Oxaliplatin for pretreated patients with advanced or metastatic pancreatic cancer: a multicenter phase II study. Cancer Invest. 2005;23(1):9-12. PMID 15779862
- [Background] HEIDELBERGER C, PARSONS DG, REMY DC. SYNTHESES OF 5-TRIFLUOROMETHYLURACIL AND 5-TRIFLUOROMETHYL-2'-DEOXYURIDINE. J Med Chem. 1964 Jan;7:1-5. doi: 10.1021/jm00331a001. No abstract available. PMID 14186018
- [Background] GOTTSCHLING H, HEIDELBERGER C. FLUORINATED PYRIMIDINES. XIX. SOME BIOLOGICAL EFFECTS OF 5-TRIFLUOROMETHYLURACIL AND 5-TRIFLUOROMETHYL-2'-DEOXYURIDINE ON ESCHERICHIA COLI AND BACTERIOPHAGE T4B. J Mol Biol. 1963 Nov;7:541-60. doi: 10.1016/s0022-2836(63)80101-1. No abstract available. PMID 14079593
- [Background] Reyes P, Heidelberger C. Fluorinated pyrimidines. XXVI. Mammalian thymidylate synthetase: its mechanism of action and inhibition by fluorinated nucleotides. Mol Pharmacol. 1965 Jul;1(1):14-30. No abstract available. PMID 4220791
- [Background] HEIDELBERGER C, ANDERSON SW. FLUORINATED PYRIMIDINES. XXI. THE TUMOR-INHIBITORY ACTIVITY OF 5-TRIFLUOROMETHYL-2'-DEOXYURIDINE. Cancer Res. 1964 Dec;24:1979-85. No abstract available. PMID 14247510
- [Background] HEIDELBERGER C, BOOHAR J, KAMPSCHROER B. FLUORINATED PYRIMIDINES. XXIV. IN VIVO METABOLISM OF 5-TRIFLUOROMETHYLURACIL-2-C-14 AND 5-TRIFLUOROMETHYL-2'-DEOXYURIDINE-2-C-14. Cancer Res. 1965 Apr;25:377-81. No abstract available. PMID 14281103
- [Background] Santi DV, Sakai TT. Thymidylate synthetase. Model studies of inhibition by 5-trifluoromethyl-2'-deoxyuridylic acid. Biochemistry. 1971 Sep 14;10(19):3598-607. doi: 10.1021/bi00795a018. No abstract available. PMID 5146573
- [Background] Fujiwara Y, Oki T, Heidelberger C. Fluorinated pyrimidines. XXXVII. Effects of 5-trifluoromethyl-2'-deoxyuridine on the synthesis of deoxyribonucleic acid of mammalian cells in culture. Mol Pharmacol. 1970 May;6(3):273-80. No abstract available. PMID 5462680
- [Background] Fujiwara Y, Heidelberger C. Fluorinated pyrimidines. 38. The incorporation of 5-trifluoromethyl-2'-deoxyuridine into the deoxyribonucleic acid of vaccinia virus. Mol Pharmacol. 1970 May;6(3):281-91. No abstract available. PMID 5443533
- [Background] Emura T, Suzuki N, Yamaguchi M, Ohshimo H, Fukushima M. A novel combination antimetabolite, TAS-102, exhibits antitumor activity in FU-resistant human cancer cells through a mechanism involving FTD incorporation in DNA. Int J Oncol. 2004 Sep;25(3):571-8. PMID 15289858
- [Background] Murakami Y, Kazuno H, Emura T, Tsujimoto H, Suzuki N, Fukushima M. Different mechanisms of acquired resistance to fluorinated pyrimidines in human colorectal cancer cells. Int J Oncol. 2000 Aug;17(2):277-83. doi: 10.3892/ijo.17.2.277. PMID 10891536
- [Background] Emura T, Suzuki N, Fujioka A, Ohshimo H, Fukushima M. Potentiation of the antitumor activity of alpha, alpha, alpha-trifluorothymidine by the co-administration of an inhibitor of thymidine phosphorylase at a suitable molar ratio in vivo. Int J Oncol. 2005 Aug;27(2):449-55. PMID 16010427
- [Background] Emura T, Murakami Y, Nakagawa F, Fukushima M, Kitazato K. A novel antimetabolite, TAS-102 retains its effect on FU-related resistant cancer cells. Int J Mol Med. 2004 Apr;13(4):545-9. PMID 15010854
- [Background] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050
- [Background] Shitara K, Doi T, Dvorkin M, Mansoor W, Arkenau HT, Prokharau A, Alsina M, Ghidini M, Faustino C, Gorbunova V, Zhavrid E, Nishikawa K, Hosokawa A, Yalcin S, Fujitani K, Beretta GD, Cutsem EV, Winkler RE, Makris L, Ilson DH, Tabernero J. Trifluridine/tipiracil versus placebo in patients with heavily pretreated metastatic gastric cancer (TAGS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1437-1448. doi: 10.1016/S1470-2045(18)30739-3. Epub 2018 Oct 21. PMID 30355453
- [Background] Overman MJ, Kopetz S, Varadhachary G, Fukushima M, Kuwata K, Mita A, Wolff RA, Hoff P, Xiong H, Abbruzzese JL. Phase I clinical study of three times a day oral administration of TAS-102 in patients with solid tumors. Cancer Invest. 2008 Oct;26(8):794-9. doi: 10.1080/07357900802087242. PMID 18798063
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Osoba D, Bezjak A, Brundage M, Zee B, Tu D, Pater J; Quality of Life Committee of the NCIC CTG. Analysis and interpretation of health-related quality-of-life data from clinical trials: basic approach of The National Cancer Institute of Canada Clinical Trials Group. Eur J Cancer. 2005 Jan;41(2):280-7. doi: 10.1016/j.ejca.2004.10.017. PMID 15661554

DOCUMENTS (1):
  • Study Protocol (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT04923529/Prot_001.pdf